CLINICAL TRIAL: NCT01752387
Title: A Study, Based on Medical Record and Questionnaire, Investigate the Management of Sportsman's Groin Hernia in Professional and Amateur Soccer Players -Results of the Follow-up in Our Department and a Comparison the Medical Literature
Brief Title: The Management of Sportsman's Groin Hernia in Professional and Amateur Soccer Players
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: EMC-0133-12
Record Dates: First submitted 2012-12-02; First posted 2012-12-19 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2012-11

CONDITIONS: Sportsman's Groin Hernia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the surgical treatment for sportsman's hernia in our department to the current literature. Our hypothesis is that combined solution for the two major problems that cause pain in this syndrome - repair the weakness in the posterior wall of the inguinal canal with "tension free" technique (mesh repair) and reducing the muscle strain on the abdominal wall by cutting, partially, the tendon of the external oblique muscle, will shorten the time to return to full physical activity in soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players who reffered to our clinic
* soccer players diagnosed with sportsman's hernia
* Failure of conservative treatment
* Underwent conventional surgery for sportsman's hernia in our department
* Completed the follow-up in our clinic
* age : 14-40
* male and female

Exclusion Criteria:

* soccer players who were diagnosed of had there surgery in other places
* soccer players who recover after conservative treatment

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: soccer players with groin pain
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2006-06; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
time to return to full physical activity | 2 month

SECONDARY OUTCOMES:
pain after the surgery | 1 week, 2 weeks and 4-6 month